CLINICAL TRIAL: NCT02529449
Title: A Phase 2, Clinical Pharmacological Study of ASP1941 in Japanese Patients With Type 1 Diabetes Mellitus
Brief Title: Pharmacodynamics, Pharmacokinetics, and Safety of ASP1941 in Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1941-CL-6001
Record Dates: First submitted 2015-08-18; First posted 2015-08-20 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: ASP1941; type 1 diabetes mellitus; SGLT2 inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — ipragliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): once daily
  Interventions: Drug: Placebo
- ASP1941 Low dose group (Experimental): once daily
  Interventions: Drug: ASP1941
- ASP1941 Middle dose group (Experimental): once daily
  Interventions: Drug: ASP1941
- ASP1941 High dose group (Experimental): once daily
  Interventions: Drug: ASP1941

INTERVENTIONS:
Drug: Placebo — Oral
  Arms: Placebo
Drug: ASP1941 — Oral
  Other Names: Suglat; Ipragliflozin
  Arms: ASP1941 High dose group; ASP1941 Low dose group; ASP1941 Middle dose group

SUMMARY:
The objective of this study is to assess pharmacodynamics, pharmacokinetics, and safety of ASP1941 in patients with type 1 diabetes mellitus when administered once daily (q.d.) for 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

At the time of obtaining informed consent:

* Subject is diagnosed with type 1 diabetes mellitus and has been treated with insulin therapy for at least 52 weeks (364 days).
* Subject is able to be admitted to the site as scheduled.
* Subject is able to record in Patient's diary from the first study drug dose in observation period until the day before the end of post observation.

At screening period:

* Subject has an HbA1c (NGSP) value of between 7.5% and 10.0%. If subject has an HbA1c value of between 7.3% and 10.2% (out of the reference range), HbA1c may be re-measured only once within the allowance range in screening period. Re-measured HbA1c (NGSP) value will be adopted for the determination.
* Subject has been receiving insulin therapy at daily doses (instructed by a doctor) within a ±20% range for at least 12weeks (83days) prior to the start of screening.
* Subject has a fasting serum C-peptide level ≤0.5 ng/mL at screening.
* Subject receives treatments for complications (except for transient diseases such as a cold) that, in the investigator's or sub-investigator's opinion, need not to be changed during the period from the start of screening to the end of the treatment period.
* Subject has body mass index (BMI) value of 20.0 to 35.0 kg/m2 at screening.

Exclusion Criteria:

At the time of obtaining informed consent:

* Subject has type 2 diabetes mellitus.
* Subject has participated or has been participating in a clinical study or a post marketing study of another drug or medical equipment within 12 weeks (84 days) prior to obtaining informed consent.
* Subject has received ASP1941 (ipragliflozin) with the exception of placebo.

At screening period:

* Subject has proliferative retinopathy (subjects with stable condition after photocoagulation etc. may be enrolled in the study).
* Subject has developed hypoglycemia unawareness (requires help of a third person) or severe hypoglycemia (diabetic coma, precoma, or convulsion) within 12 weeks (84 days) prior to the start of screening.
* Subject has developed diabetic ketoacidosis within 12 weeks (84 days) prior to the start of screening.
* Subject has chronic disease(s) which require the continuous use of corticosteroids or immunosuppressants (oral administration, injection, inhalation, or suppository).
* Subject has received hypoglycemic agent(s) other than insulin within 12 weeks (83 days) prior to the start of screening.
* Subject with perioperative, severe infection or serious injury.
* Subject whose serum creatinine value exceeds the upper limit of normal range at screening.
* Subject has a urinary albumin/urinary creatinine ratio>300 mg/g in urinalysis at screening.
* Subject has a history of clinically significant renal disease(s) such as renovascular occlusive disease, nephrectomy, and/or renal transplant.
* Subject has AST and ALT >2 ×ULN or T-Bil >1.5 × ULN at screening, or has a history of serious hepatic diseases.
* Subject presents with symptoms of dysuria, anuria, oliguria and urinary retention.
* Subject has a history of recurrent urinary tract infections and recurrent genital infections (developed 3 times or more within 24 weeks (168 days) prior to the start of screening).
* Subject has urinary tract infection or genital infection with subjective symptoms.
* Subject has a history of angina unstable, myocardial infarction, angioplasty, and serious heart disease (NYHA Class II-IV) within 24 weeks (168 days) prior to the start of screening, or has complications of heart disease that, in the investigator's or sub-investigator's opinion, may interfere with the evaluation of safety of ASP1941.
* Subject has uncontrolled blood pressure (systolic blood pressure≥160 mmHg or diastolic blood pressure≥100 mmHg in the supine position after a 5-minute rest at screening ).
* Subject has serious gastrointestinal disease or a history of serious gastrointestinal operation.
* Subject has malignant tumors concomitantly (subject may be enrolled in the study if the subject has a history of a malignant tumor which has not recurred without any treatment within 5 years prior to the start of screening).
* Subject has psychiatric disorder that makes the subject unsuitable for study participation.
* Subject has drug addiction or alcohol abuse.
* Subject has a history of drug allergies.
* Subject is unable to adhere to any of the compliance such as hospital visits and dose instruction specified in this study, or does not agree with it.
* Subject has donated 400 mL of whole blood within 90 days, 200 mL of whole blood within 30 days, or blood components within 14 days prior to the start of screening.
* Subject has any condition that, in the investigator's or sub-investigator's opinion, makes the subject unsuitable for study participation.

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-03-19 (Actual); Study Completion 2016-03-19 (Actual)

PRIMARY OUTCOMES:
Daily profile of plasma glucose levels | up to Day 14
Area under the concentration-time curve (AUC) 0-24hr (AUC0-24h) of plasma glucose levels | at Day -1, Day 1 and Day 14
AUC0-3h of plasma glucose levels | at Day -1, Day 1 and Day 14
AUC0-4h of plasma glucose levels | up to Day 14
AUC0-10h of plasma glucose levels | up to Day 14
Fasting plasma glucose levels | up to Day 21
Glycoalbumin | up to Day 21
Urinary glucose excretion | up to Day 14
Urinary glucose excretion rate | up to Day 14
Urine volume | up to Day 14
Urinary glucose concentration | up to Day 15
Body weight | up to Day 21
Renal glucose clearance | up to Day 14
Plasma concentration of unchanged ASP1941 | up to Day 14
Urinary concentration of unchanged ASP1941 | up to Day 14
Pharmacokinetics (PK) parameter of ASP1941 in plasma: AUC from time 0 extrapolated to infinity (AUCinf) | at Day 1
PK parameter of ASP1941 in plasma: AUC from the time of dosing to the last measurable concentration (AUClast) | at Day 1 and Day 14
PK parameter of ASP1941 in plasma: AUC from the time of dosing to 24 hr (AUC0-24h) | at Day 1 and Day 14
PK parameter of ASP1941 in plasma: Oral Clearance (CL/F) | at Day 1 and Day 14
PK parameter of ASP1941 in plasma: Maximum concentration (Cmax) | at Day 1 and Day 14
PK parameter of ASP1941 in plasma: Terminal Elimination Half-life (t1/2) | at Day 1 and Day 14
PK parameter of ASP1941 in plasma: Time of the Maximum Concentration (tmax) | at Day 1 and Day 14
PK parameter of ASP1941 in urine: Amount excreted in urine between time (Ae) | at Day 1 and Day 14
PK parameter of ASP1941 in urine: % of the dose of excreted in urine (Ae%) | at Day 1 and Day 14
PK parameter of ASP1941 in plasma and urine: Renal Clearance (CLr) | at Day 1 and Day 14
Safety assessed by vital signs | up to Day 21
  Supine blood pressure and supine pulse rate
Safety assessed by 12-lead electrocardiogram | up to Day 21
Safety assessed by laboratory tests | up to Day 21
  Hematology, biochemistry and urinalysis
Safety assessed by self-monitored blood glucose levels | up to Day 21
Safety assessed by Adverse events | up to Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (11):
- Japan (11):
  - Site JP00006, Aichi
  - Site JP00002, Fukuoka
  - Site JP00009, Gunma
  - Site JP00001, Ibaraki
  - Site JP00005, Kanagawa
  - Site JP00008, Kanagawa
  - Site JP00003, Okayama
  - Site JP00004, Osaka
  - Site JP00010, Osaka
  - Site JP00011, Osaka
  - Site JP00007, Tokyo

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Toyoshima J, Saito M, Kaibara A, Isaka H, Sakatani T. Comparison of the Pharmacokinetic and Pharmacodynamic Relationship of Ipragliflozin Between Patients With Type 1 and Type 2 Diabetes Mellitus. Clin Ther. 2020 Sep;42(9):1787-1798.e3. doi: 10.1016/j.clinthera.2020.07.009. Epub 2020 Aug 21. PMID 32839028
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/hcp/study.aspx?ID=307